CLINICAL TRIAL: NCT06905938
Title: Comparison of the Clinical Outcomes of Extended Depth of Focus Intraocular Lenses and Monofocal Intraocular Lenses in Patients With High Myopia Undergoing Cataract Surgery.
Brief Title: Comparing Monofocal IOLs in Highly Myopic Cataract Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Other Study IDs: H2025-014-K-13
Record Dates: First submitted 2025-03-12; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ICB00 implantation after cataract surgery.: Undergoing micro-incision cataract surgery with the implantation of an extended depth of focus (EDOF) intraocular lens (ICB).
  Interventions: Other: no intervention
- ZCB00 implantation after cataract surgery.: Performing micro-incision cataract surgery and implanting a ZCB (presumably an abbreviation specific to a certain type of intraocular lens) intraocular lens
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Comparison of Postoperative Outcomes in Patients with High Myopia Undergoing Cataract Surgery Implanted with Extended Depth of Focus Intraocular Lens (ICB00) and Monofocal Intraocular Lens (ZCB00)

DETAILED DESCRIPTION:
In this study, we aim to compare the visual outcomes and quality of life between highly myopic patients with cataracts who receive implantation of extended depth of focus (EDOF) intraocular lenses (ICB00) and monofocal intraocular lenses (ZCB00). This is a case-control study, planning to recruit 64 highly myopic patients with cataracts, aged between 40 and 70, with 32 in each group. The primary endpoints of the study are the best-corrected visual acuity (BCVA) and defocus curve at 6 months postoperatively. Secondary endpoints include uncorrected visual acuity (UCVA), contrast sensitivity, intraocular pressure, and assessments of patient satisfaction and quality of life. These will be evaluated using standardized questionnaires such as the VF-14, the PRSIQ spectacle dependency scale, and reading speed tests to quantify changes in vision-related quality of life. Patients will undergo comprehensive ophthalmic examinations preoperatively and at 6 months postoperatively, including slit-lamp anterior segment examination, fundus examination, corneal topography, and intraocular pressure testing. Additionally, questionnaires will be used to assess patients' subjective satisfaction with visual improvement and spectacle needs in daily life. All data will be statistically analyzed to compare the effects of the two types of intraocular lenses. Continuous variables will be analyzed using t-tests or Mann-Whitney U tests, and categorical variables will be analyzed using chi-square tests. The level of statistical significance is set at p<0.05. Through this study, we hope to determine whether the use of EDOF intraocular lenses provides better visual outcomes and quality of life compared to monofocal intraocular lenses in highly myopic patients with cataracts. The results of this study will provide a more scientific basis for the choice of intraocular lenses in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* 1: The patients are between 40 and 70 years old.

  2: Ocular axis > 26mm

  3: Able to understand, cooperate and complete all follow-up.

Exclusion Criteria:

* 1: Moderate and severe dry eye

  2: There is macular degeneration complicated by high myopia.

  3: Combined with other ophthalmic diseases

  4: Previous history of ophthalmic surgery.

  5: There are intraoperative or postoperative complications.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Included in Eye Hospital of Wenzhou Medical University for "phacoemulsification combined with intraocular lens implantation"
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Defocus curve | Three months after operation
  On the basis of BCDVA, add +2.5~-5.0D spherical lenses (decreasing at intervals of 0.5D) before the patient's operation, record the logMAR vision of the patient at each added spherical lens degree, and draw the average Defocus Curve with the added spherical lens degree as the abscissa and the average vision of each corresponding degree as the ordinate.
Far, middle and near vision | Three months after operation
  The naked eye vision was measured at 5m, 70cm and 40cm respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Yune, Principal Investigator — Ethics Committee of the affiliated Ophthalmology Hospital of Wenzhou Medical University
Locations (1):
- Ophthalmology and Optometry Hos, Hanzhou, Zhejian, China

IPD SHARING:
Plan to Share IPD: No